CLINICAL TRIAL: NCT05731739
Title: A Retrospective Analysis of Clinical Outcomes of IV Lidocaine Infusion for Neuropathic Pain: Assessing Predictors of Clinically Relevant Analgesia and to Report the Efficacy and Side Effect Profile of Infusion
Brief Title: IV Lidocaine Infusion for Neuropathic Pain
Status: Withdrawn | Type: Observational
Why Stopped: Resources did not come to fruition
Sponsor: Henry Ford Health System (Other)
Responsible Party: Principal Investigator, Gaurav Chauhan, RESIDENT ANESTHESIOLOGY, Henry Ford Health System
Other Study IDs: HFHS PAIN MEDICINE
Record Dates: First submitted 2016-04-06; First posted 2023-02-16 (Actual); Last update posted 2023-02-16 (Actual); Status verified 2023-02

CONDITIONS: Neuropathic Pain; Complex Regional Pain Syndrome; Chronic Pain
Keywords: LIDOCAINE, NEUROPATHIC PAIN, CHRONIC PAIN
MeSH Terms: conditions — Neuralgia; Complex Regional Pain Syndromes; Chronic Pain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- RESPONDERS: The investigators will define responders as patients achieving Numerical Rating Score (NRS) reductions of 30% or greater based on literature defined criteria for meaningful reductions in pain scores
- NON RESPONDERS: When a patient failed to respond to the lidocaine infusion, they were given the option to have repeat infusion after four weeks. If no response was obtained, despite two infusions, this was considered as a failure of treatment and no further lidocaine infusions were conducted. Patient will be labelled as a non responder

SUMMARY:
The investigators will conduct a retrospective cohort study of patients who have undergone i.v. lidocaine infusions in the previous 2 years for suspected neuropathic pain of heterogeneous origin. The investigators hypothesize that the analgesic response to intravenous (i.v.) lidocaine will be bimodal with clear responders and clear non-responders. The investigators also hypothesize that more refractory patients, who have failed previous multimodal analgesic therapy, will be less likely to respond to i.v. lidocaine. The investigators goals are to report what percentage of patients will achieve relief, the degree of relief that can be expected, and identify the type of patients who will most likely to benefit from systemic lidocaine. The investigators secondary objective is to report the correlation between infusion rates and patterns of infusion rate adjustments with regard to efficacy and adverse effects.

DETAILED DESCRIPTION:
HYPOTHESIS On the basis of investigators' clinical experience, The investigators hypothesize that the analgesic response to intravenous (i.v.) lidocaine will be bimodal with clear responders and clear non-responders. The investigators also hypothesize that more refractory patients, specifically patients with pain of longer duration and patients who have failed previous multimodal analgesic therapy, will be less likely to respond to i.v. lidocaine. To test the hypotheses, we will identify the distribution of pain relief in the enrolled cohort. The investigators will define responders as patients achieving Numerical Rating Score (NRS) reductions of 30% or greater based on literature defined criteria for meaningful reductions in pain scores.The investigators goals are to report what proportion of patients will achieve relief, the degree of relief that can be expected, and identify the type of patients who will most likely to benefit from systemic lidocaine. The investigators also hypothesize that degree of pain relief in a responder to i.v. lidocaine will be translated in the form of concomitant decrease in quantitative measures of PHQ-9 scales and Oswestry index scales. The investigators secondary objective is to report the correlation between infusion rates and patterns of infusion rate adjustments with regard to efficacy and adverse effects.

DESIGN AND SETTING The investigators will conduct a retrospective cohort study of patients who have undergone IV lidocaine infusions for suspected neuropathic pain. All patients will be recruited from the Pain Management Clinic at Henry Ford Health System.

STUDY PARTICIPANTS The investigators will secure approval from the Institutional Review Board and ethics committee of the institution. The investigators will review patients' information and their treatment data through the electronic medical record (EPIC) of the pain management clinic. The investigators will screen sequential charts of previous two years to identify patients who have undergone i.v. lidocaine infusions for Neuropathic Pain of heterogeneous origin. Inclusion criteria will include: neuropathic pain suspected by the board certified pain specialist assessing the patient based on the presence of allodynia, hyperalgesia, hyperpathia and hyperesthesia or hypesthesia. The exclusion criteria will include patients that refused subsequent i.v. lidocaine infusions or were lost to follow up.

DATA COLLECTION AND INDEPENDENT VARIABLES Independent variables examined will include the patient's age, sex, body mass index, indication, duration of pain problem, dates of treatment, dose, infusion time, adverse events, action taken as a result of an adverse event, duration of treatment, reason for discontinuation, pre and post infusion NRSs of pain, vital signs that were taken pre-infusion, during infusion and post-infusion, previous trials of alternative pain medication and current or previous substance abuse.

STATISTICAL ANALYSIS Initial analysis of patient's age, sex, pain severity, pain duration, number alternative medication tried, with comparison between lidocaine responders and non-responders will be done using Student t test or χ2 test as appropriate. All statistical tests will be 2-sided. A p value less than 0.05 will be considered statistically significant. Normality of data will be assessed with Kolmogorov-Smirnov test. Odds ratios with 95% confidence intervals (CIs) will be calculated. SAS version 9.4 (SAS Institute, Cary, NC) will be used for all analysis.

ELIGIBILITY:
Inclusion Criteria:

* patient with neuropathic pain
* patient enrolled for lidocaine infusion

Exclusion Criteria:

* refusal to consent
* lost to follow-up

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients' information and their treatment data will be identified through the electronic medical record (EPIC) of the pain management clinic. The investigators will screen sequential charts of previous two years to identify patients who have undergone i.v. lidocaine infusions for Neuropathic Pain of heterogeneous origin (e.g., post-herpetic neuralgia, post surgical nerve injury, lumbar radiculopathy).
  Inclusion criteria will include: neuropathic pain suspected by the board certified pain specialist assessing the patient based on the presence of allodynia, hyperalgesia, hyperpathia and hyperesthesia or hypesthesia.
  The exclusion criteria will include patients that refused subsequent i.v. lidocaine infusions or were lost to follow up.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2016-04; Primary Completion 2023-01 (Actual); Study Completion 2023-01 (Actual)

PRIMARY OUTCOMES:
Identify the type of patients who will most likely to benefit from systemic lidocaine. | April, 2016 - August, 2016
  Primary aim is to test the hypothesis that the analgesic response to intravenous (i.v.) lidocaine are bimodal with responders and non-responders.

SECONDARY OUTCOMES:
Quantify the efficacy of lidocaine infusion in terms of duration of meaningful decrease in pain in patients with neuropathic pain | April, 2016 - August, 2016
  secondary goals are to report what proportion of patients will achieve clinically meaningful relief, which is defined as >50% reduction in the baseline numeric rating pain score.
Our last objective is to report the adverse effects | April, 2016 - August, 2016
  Will recored recognized side effects (tinnitus, perioral numbnes, dysarthria etc.) which used as a basis for titrating the therapy to minimal effective dose

CONTACTS AND LOCATIONS:
Overall Officials: NABIL SIBAI, M.D., Study Chair — HENRY FORD HEALTH SYSTEMS
Locations (1):
- Henry Ford Health Systems, Detroit, Michigan, United States

IPD SHARING:
Plan to Share IPD: No